CLINICAL TRIAL: NCT01983800
Title: Use of Volatile Anesthetics for Long-Term Sedation In Critically Ill Patients
Brief Title: AnaConDa Long Term Sedation Study
Acronym: VALTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHN 13-5845
Record Dates: First submitted 2013-07-02; First posted 2013-11-14 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2020-05

CONDITIONS: Intubated Requiring Sedation for Greater Than 48 Hours
Keywords: Mechanical Ventilation; Volatile Sedation; Intravenous Sedation; Delirium
MeSH Terms: conditions — Delirium | interventions — Isoflurane; Propofol; Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intravenous propofol/midazolam (Active Comparator): Sedation using intravenous propofol/midazolam, sedation will be titrated to a Riker Agitation Sedation Score
  Interventions: Drug: Propofol/midazolam
- isoflurane (Active Comparator): Sedation using inhaled isoflurane, sedation will be titrated to a Riker Agitation Sedation Score
  Interventions: Drug: Isoflurane

INTERVENTIONS:
Drug: Isoflurane
  Arms: isoflurane
Drug: Propofol/midazolam
  Arms: intravenous propofol/midazolam

SUMMARY:
Heavy sedation or sleep is a common problem within the intensive care unit (ICU) using our standard intravenous medications. This commonly leads to confusion, low blood pressure, slow wake up and removal of the artificial breathing tube (extubation), which prolongs ICU stay. Using inhaled volatile anesthetic agents are likely to improve these patient outcomes. This unique project is the first North American study looking at using volatiles for patients who need longer-term ICU sedation. This project has excellent potential at lowering these complications and improving quality of care, which will lower patient ICU stay and healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* adult ICU patients expected to be ventilated > 48 hours

Exclusion Criteria:

* age < 18 years
* history of malignant hyperthermia
* propofol infusion syndrome
* evidence of raised intracranial pressure
* 6-month mortality risk from pre-existing condition > 50%
* lack of commitment to maximal treatment
* pregnant
* NebulizedFlolan
* tidal volume <350ml
* patients on one lung ventilation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
atmospheric volatile concentration | daily
  Daily assessment of atmospheric volatile levels will be measured using photometric multigas infrared analyzer
Sedation | daily
  adherence to the volatile sedation, sedation will be guided by explicit protocols targeting a Sedation-Agitation Score (SAS) of 3-4
Feasibility | 2 years
  assess rate of patient recruitment and barriers to recruitment
Education Tool | 2 years
  multidisciplinary feedback regarding teaching package, protocol, quality of sedation
serum fluoride levels | every 2 days
  Measurements will be taken 24 hours post sedation and every 2 days until while on sedation followed by 2 further samples after discontinuation of sedation.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Jerath, MD, Principal Investigator — Toronto General Hospital, University Health Network
Locations (2):
- Canada (2):
  - Ottawa Heart Institute, Ottawa, Ontario
  - Toronto General Hospital, University Health Network, Toronto, Ontario

REFERENCES:
- [Derived] Jerath A, Ferguson ND, Steel A, Wijeysundera D, Macdonald J, Wasowicz M. The use of volatile anesthetic agents for long-term critical care sedation (VALTS): study protocol for a pilot randomized controlled trial. Trials. 2015 Dec 9;16:560. doi: 10.1186/s13063-015-1083-5. PMID 26646404